CLINICAL TRIAL: NCT05679102
Title: Effect of Atorvastatin in the Management of Hypertension
Brief Title: Atorvastatin as an Antihypertensive Agent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Himayat Ullah (Other)
Collaborators: Ayub Teaching Hospital (Other); Khyber Medical University Peshawar (Other)
Responsible Party: Sponsor-Investigator, Himayat Ullah, Assistant Professor, Shaqra University
Organization: Shaqra University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIR/KMU-EB/EA/000560
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Atorvastatin Antihypertensive Effect
MeSH Terms: interventions — Amlodipine; Tablets; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amlopdipine only (Active Comparator): Newly diagnosed hypertensive patients who will be given only amlodipine.
  Interventions: Drug: Amlodipine 5 MG Oral Tablet
- Amlodipine and Atorvastatin (Active Comparator): Newly diagnosed hypertensive patients who will be given Amlodipine and Atorvastatin.
  Interventions: Drug: Amlodipine 5 MG / Atorvastatin 10 MG Oral Tablet

INTERVENTIONS:
Drug: Amlodipine 5 MG Oral Tablet — one group will be given only Amlodipine 5MG once daily
  Arms: Amlopdipine only
Drug: Amlodipine 5 MG / Atorvastatin 10 MG Oral Tablet — one group will be given Amlodipine 5mg plus Atorvastatin 10MG once daily
  Arms: Amlodipine and Atorvastatin

SUMMARY:
This study is aimed to see the antihypertensive effect of statin (Atorvastatin) as certain animal models have shown that statins have the voltage-gated calcium channel blocking effect. It will be a randomized controlled trial that will be done in Ayub Hospital Complex Abbottabad. After ethical approval, 120 patients with newly diagnosed hypertension belonging to either gender and aged 35 and above will be enrolled in the trial. They will randomly be grouped into two groups with each group comprising 60 patients. One group will be administered Amlodipine 5 mg PO once a day, while the other one will be given 5mg Amlodipine plus 10 mg Atorvastatin. The patients will be examined on a follow-up visit 14 days later and blood pressure will be recorded as per protocols.

ELIGIBILITY:
Inclusion Criteria:

- The inclusion criteria for the study were all newly diagnosed hypertensive patients aged 35 years and above with normal lipid profile

Exclusion Criteria:

* Patients with a history of dyslipidemias, diabetes mellites, chronic kidney disease, and ischemic heart disease

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Antihypertensive effect of atorvastatin | 14 days
  patients receiving atorvastatin based combination should have more decrease in the blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Shaqra University, Shaqra, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
IPD will be available to the principle researcher and corresponding researcher only.